## Appendix D: Statement of consent

Regarding "Transmission blocking malaria vaccine R0.6C (STOP-TRANS)"

I have read the information letter. The study has been explained to me and I had the chance to ask questions. I had enough time to decide whether to participate. I know that participation is voluntary. I also know that I can decide at any time to withdraw my participation in the study. I don't have to disclose my reason to stop.

By signing this statement, I agree to take part in this study. Furthermore:

- I give permission to the researcher to inform my general practitioner that I am participating in this study.
- I give permission to the researcher to request information from my GP about my medical history or medication use if necessary.
- I give permission to the researcher to provide my GP or specialist with information about unexpected findings in the study that are important for my health.
- I give permission to the researchers to collect and use my data and blood samples. The
  researchers will only do this to answer the research question of this study. And to register the
  drug.
- I know that some people will be able to view all of my data for the verification of the study.
   Those people are described in this information letter. I give these people permission to view my data for this purpose.
- I know that I cannot get pregnant during the study. The researcher has discussed acceptable contraception methods with me.
- I give permission to transfer my data and blood samples to countries outside the European Union where the European guidelines for the protection of personal data may not apply. The data and blood samples must be transferred encrypted and without my name.
- Please tick yes or no in the table below:

| I give permission to store my data and (remaining) blood samples in order to use it | Yes | No |
|---|---|---|
| for other research, as stated in the information letter. The human material is stored | | |
| for 15 years for this purpose. | | |
| Name (subject): | | |
| Signature: Date : / / | | |
| I declare that I have fully informed this subject about the study. If any information be known during the study that could influence the subject's consent, I will let this test sknow in time. Name (researcher or representatieve): | | |
| The subject will receive a complete information letter, together with a signed version | of the | |

consent form.